CLINICAL TRIAL: NCT06579937
Title: Esketamine for the Prevention of Postoperative Behavioral Changes in Children Undergoing Tonsillectomy and/or Adenoidectomy: a Randomized Controlled Trial
Brief Title: Effects of Esketamine on Postoperative Behavioral Changes in Children Undergoing Tonsillectomy and/or Adenoidectomy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Clinical Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K2023-02-005
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Behavior Problem
Keywords: esketamine; postoperative negative behavioral change; pediatrics; emergence delirium; tonsillectomy; adenoidectomy
MeSH Terms: conditions — Mental Disorders; Emergence Delirium | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esketamine group (Experimental): During anesthesia induction, 0.2 mg/kg esketamine was administered intravenously.
  Interventions: Drug: Esketamine hydrochloride
- Control group (Placebo Comparator): During anesthesia induction, an equal volume of 0.9% saline was administered intravenously.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine hydrochloride — During anesthesia induction, a 0.2 mg/kg esketamine bolus was administered intravenously.
  Other Names: esketamine hydrochloride injection
  Arms: Esketamine group
Drug: normal saline — During anesthesia induction, a bolus of equal 0.9% saline was administered intravenously.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn the effect of intravenous esketamine in postoperative negative behavior changes in children compared to placebo (a look-alike substance that contains no drug). It will also learn about the effect of esketamine in emergence delirium. The main questions are:

Dose esketamine lower the incidence of postoperative negative behavior changes compared to placebo? Dose esketamine lower the incidence of emergence delirium compared to placebo? Researchers will compare esketamine to placebo to see if esketamine works to treat postoperative negative behavior change and emergence delirium.

Participants will:

Receive intravenous esketamine or placebo (a look-alike substance that contains no drug) during anesthesia induction; Fill in the Post hospitalization behavior questionnaire for ambulatory surgery postoperative 1, 7, and 30

DETAILED DESCRIPTION:
Approximately half of children who undergo general anesthesia experience emergence delirium (ED) and postoperative negative behavioral changes (PNBC). There was a positive correlation between delirium during recovery and the change in negative behaviour after the operation.

Esketamine has sedative, analgesic and anti-traumatic stress effects. Based on literature analysis and preliminary trials, this study suggests that intraoperative use of low-dose esketamine may reduce the incidence of emergence delirium and postoperative negative behavior changes in children.

This prospective randomized controlled trial was conducted to compare the effect of intravenous esketamine in the incidence of emergence delirium and postoperative negative behavior changes in children compared to placebo (a look-alike substance that contains no drug) to provide a reference for optimizing clinical anesthesia medication regimens.

ELIGIBILITY:
Inclusion Criteria:

* American society of Aneshesiologists physical status I or II;
* Aged 3-7 years;
* Scheduled for elective tonsillectomy and (or) adenoidectomy.

Exclusion Criteria:

* Parents refusing to allow their children to participate;
* Intake of sedative or analgesic medication within 48 hours before surgery;
* Developmental delay;
* Psychosis;
* Body mass index > 30 kg/m2;
* Allergy to study drugs;
* Major life changes 1 month before the operation, such as the divorce of parents, death of parents, moving to a new home, changing to a new kindergarten, etc.;
* Any other conditions that precluded study inclusion.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Estimated)
Dates: Start 2024-09-02 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative negative behavior changes | Postoperative day 7
  Postoperative negative behavior changes were assessed with Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).

SECONDARY OUTCOMES:
Incidence of postoperative negative behavior changes | Postoperative day 1
  Postoperative negative behavior changes were assessed with Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).
Incidence of emergence delirium | Within 30 minutes after extubation
  Emergence delirium was assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale (defined as a PAED score of ≥10).
Incidence of postoperative negative behavior changes | Postoperative day 30
  Postoperative negative behavior changes were assessed with Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).
Postoperative pain intensity | Within 30 minutes after extubation
  Postoperative pain intensity will be measured using the face, legs, activity, cry, and consolability scale.
Preoperative anxiety | Before the intervention in holding area
  Preoperative anxiety will be assessed using the modified Yale preoperative anxiety scale. Scores range from 23 to 100 with higher scores indicating greater anxiety.
Emergence time | About up to 30 minutes postoperatively
  Emergence time is defined as the interval from discontinuation of inhalation anesthetic to eye-opening on verbal command.
Parental satisfaction | Postoperative day 1
  Parental satisfaction is self-reported using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Length of postanesthesia care unit stay | Up to 60 minutes postoperatively
  Length of postanesthesia care unit (PACU) stay is defined as the time between arrival in the PACU and readiness for discharge from the PACU (defined as a modified Aldrete score of ≥9).
Incidence of adverse events | Up to 24 hours postoperatively
  Adverse events such as bradycardia, tachycardia, hypertension, hypotension, and hypoxia will be recorded during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD, Study Chair — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the individual deidentified participant data underlying published results, the study protocol, and the statistical analysis plan can be accessed upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The researcher would like to share the individual deidentified participant data beginning three months following the publication of the main results.
Access Criteria: All the individual participant data collected during the trial, the study protocol, the statistical analysis plan, and the clinical study report can be accessed with approval from the corresponding author.